CLINICAL TRIAL: NCT04312568
Title: Evaluate Safety, Tolerability and Pharmacokinetics of Fadanafil （XZP-5849）in Chinese Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5849-CPK-1001
Record Dates: First submitted 2020-03-11; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Healthy Subject
Keywords: Healthy Subject; PK Study; Tolerability; Safety Evaluation
MeSH Terms: interventions — 1,2-dibenzoyl-tert-butylhydrazine

STUDY DESIGN:
Intervention Model Description: 8 dose groups within 12.5mg~500mg for single dose tolerability study to carrried out from low-dose group to high dose group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fadanafil (Experimental): 8 group: 12.5mg one dose; 25mg one dose; 50mg one dose; 100mg one dose; 200mg one dose; 300mg one dose; 400mg one dose; 500mg one dose
  Interventions: Drug: Fadanafil
- Placebo (Placebo Comparator): 8 group: 12.5mg one dose; 25mg one dose; 50mg one dose; 100mg one dose; 200mg one dose; 300mg one dose; 400mg one dose; 500mg one dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fadanafil — Dose escalation for 8 groups: 12.5mg one dose, 25mg one dose, 50mg one dose, 100mg one dose, 200mg one dose, 300mg one dose, 400mg one dose, 500mg one dose
  Other Names: 5849
  Arms: Fadanafil
Drug: Placebo — Dose escalation for 8 groups: 12.5mg one dose, 25mg one dose, 50mg one dose, 100mg one dose, 200mg one dose, 300mg one dose, 400mg one dose, 500mg one dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety , tolerability, and pharmacokinetics of ascending single dose Fadanafil （XZP-5849）in Chinese healthy adult male subjects. This is the first XZP-5849 clinical study

DETAILED DESCRIPTION:
XZP-5849 is a selective phosphodiesterase (PDE5) inhibitor. The proposed randomized Phase 1 trial is a double-blind, placebo-controlled, single ascending dose study in approximately 66 Chinese healthy adult male subjects. The study consists of 8 cohorts (1 cohort per dose level). Each subject will participate in only one cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects 18-45 years old, inclusive.
* Body weight ≥50kg and Body Mass Index: 19.0~25.0 kg/m2, inclusive
* subjects should be willing to take appropriate contraceptive measures during the period of taking the study drug and within 6 months after discontinuation to avoid pregnancy of their partners.

Exclusion Criteria:

* Subjects who have a history of clinical significanct drug allergy (especially those who are known or suspected to have a history of allergy to any PDE-5 inhibitor or its components) or a history of atopic allergic diseases (asthma, urticaria, eczema dermatitis) or severe allergic constitution.
* History of clinically significant ECG abnormality or family history of long QT syndrome (grandparents, parents, brothers and sisters).
* Subjects with serious systemic diseases, such as respiratory, blood, endocrine, cardiovascular and cerebrovascular diseases or mental disorders.
* Subjects who have used over-the-counter drugs, health products, herbal medicine or traditional Chinese medicine within 2 weeks before screening, or are taking foods that affect CYP3A4, such as grapefruit or drinks containing grapefruit (except those who occasionally take paracetamol, but the total maximum dose cannot exceed 1g, and the drug is not allowed to take orally within 48 hours before the first administration).
* Subjects who have used any prescription drugs (especially CYP3A4 inhibitors, nitrates, α receptor blockers, drugs potential to cause QT interval prolongation, etc.) within 4 weeks before screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Electrocardiogram (ECG) | Change from Baseline to 1, 2,4,6,8,12,24,36,46 hours after dosing.
  To evaluate subject ECG Changing information
Pharmacokinetic Parameter AUC(0-24) | Pre dose and 0.25,0.5,0.75,1,1.5, 2, 2.5, 4, 6,8,12, 24,36 hours after Dosing
  AUC(0-24) of Fadanafile is area under the curve
Blood Pressure and Heart Rate | Change from Baseline to 1, 2,4,6,8,12,24,36,46 hours after dosing
  To evaluate subject Blood Pressure and Heart Rate Changing information

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Li, Doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Haiyan Li, Beijing, Beijing Municipality, China